Using Grassroots Wellness Coaching to Enhance Reach and Sustainability of Behavioral Weight Management

PI: Maghboeba Mosavel, PhD, Professor: (804) 628-2929 and Jessica G. LaRose, PhD, Professor: (/804) 628-7521

Both consents were approved by the IRB on 1/9/2025, the template revision date is 10/23/2024

# Permission to Take Part in a Human Research /Study

ICF version number: Version 1

Title of research study¹: Using Grassroots Wellness Coaching to Enhance Reach and Sustainability of Behavioral Weight Management

*I/nvestigator:* Maghboeba Mosavel, PhD, Professor: (804) 628-2929 and Jessica G. LaRose, PhD, Professor: (/804) 628-7521

**<u>Key Information</u>**: The following is a short summary of this study to help you decide whether or not to be a part o/f this study. More detailed information is listed later on in this form.

# Why am I being invited to take part in a research study?

We/ invite you to take part in a research study because

- You were eligible to participate in the W.E. 2.0 Project as a Wellness Ambassador, or
- You were eligible to participate in the W.E. 2.0 Project as a participant, or
- You participated and completed the 12-week program as a Wellness Ambassador or participant

# What should I know about a research study?

- Someone will explain this research study to you.
- W/hether or not you take part is up to you.
- You can choose not to take part.
- You can agree to take part and later change your mind.
- Your decision will not be held against you.
- You can ask all the questions you want before you decide.

# Why is this research being done?

You are being asked to take part in this research project because you participated in the W.E. 2.0 research study. The purpose of this project is to find out what helps or makes it harder for House Chat meetings to be successful over time. We also want to figure out the best ways to support and keep these programs going in the comm/unity.

If you agree to participate in this study, you will be asked to complete a one-time Zoom meeting with a member of the WE 2.0 Project research team. You may experience several personal benefits from taking part in this research. Sharing your experiences openly may give you a chance to reflect on your interest and or participation in the WE project, leading to personal insights.

### How long will the research last and what will I need to do?

You will be asked to participate in a one-time, 45-minute Zoom meeting to share your experience with a member of the WE research team. Only the audio portion of this meeting will be downloaded and analyzed for the results. There are no additional tasks to be completed once you finish the interview.

More detailed information about the study procedures can be found under "What happens if I say yes, I want to be in this research?"


Template Revision Date: October 23, 2024

<sup>&</sup>lt;sup>1</sup> This template satisfies AAHRPP elements I.1.G, I.4.A, I-9, II.3.C-II.3.C.1, II.3.E, II.3.F, II.4.B, III.1.F, III.1.G

# Is there any way being in this study could be bad for me?

This study is considered low risk. You won't face any physical harm or emotional distress, and we've designed everything to respect your privacy and make sure you feel comfortable and at ease throughout the process.

We do understand that sharing your experiences might feel a little uncomfortable. If that happens, we want you to know those feelings are normal and should only be short-term. To help, we'll create a supportive, judgment-free space during the interviews. This study is all about understanding your experiences—not judging your success or failure. Your privacy and comfort are our top priorities.

# Will being in this study help me in any way?

We cannot promise any benefits to you from your taking part in this research. However, possible benefits include the opportunity to share your personal experiences and to have your opinions heard and valued through self-reflection and lessons learned.

Your experiences and insights can possibly help improve the program to make it more beneficial for others in Petersburg or communities outside of Petersburg.

# What happens if I do not want to be in this research?

Participation in this research is completely voluntary. You can decide to participate, not participate, or discontinue participation at any time without penalty or loss of benefits to which you are otherwise entitled.

Your alternative to participating in this research study is to not participate.

<u>Detailed Information</u>: The following is more detailed information about this study in addition to the information listed above.

### Who can I talk to?

If you have questions, concerns, or complaints, or think the research has hurt you, talk to the research team at (804) 396-4556 or send us an email: WEPetersburg2.0@vcuhealth.org.

This research has been reviewed and approved by an Institutional Review Board ("IRB"). You may talk to them at (804) 828-0868 or HRPP@vcu.edu if:

- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.
- You want to talk to someone besides the research team.
- You have questions about your rights as a research subject.
- You want to get information or provide input about this research.

### How many people will be studied?

We expect to speak with a selected group of WE wellness ambassadors and participants and it could include up to 50 individuals.

# What happens if I say yes, I want to be in this research?

If you agree to participate in this study, you will be asked to complete a one-time, 45 minute Zoom audio meeting with a member of the WE 2.0 Project research team. This interview will be scheduled at a time that is most convenient for you.

# What are my responsibilities if I take part in this research?

During this meeting, you will be responsible for providing your personal thoughts about various aspects of the WE 2.0 and offer any suggestions that could improve this study for other communities in the future.

# What happens if I say yes, but I change my mind later?

You can leave the research at any time; it will not be held against you. If you choose to withdraw for any reason, all data collected will be carefully disposed of to eliminate any risk of personal information being misused. In addition, you will not be withdrawn from the study without your direct consent.

All data that is collected will be used for research purposes only. Your data will be identified by an ID number and safely stored in our database. Access to all data will be limited to study personnel.

We will do our best to protect your data during storage and when they are shared. However, there remains a possibility that someone could identify you. There is also the possibility that people who are not supposed to might access your data and samples. In either case, we cannot reduce the risk to zero.

# What happens to the information collected for the research?

Efforts will be made to limit the use and disclosure of your personal information, including research study records, to people who have a need to review this information. We cannot promise complete secrecy. Organizations that may inspect and copy your information include the IRB and other representatives of this organization.

# Will my data or samples be used for future research?

Your information collected as part of this research will not be used or distributed for future research studies, even if all of your identifiers are removed.

# Can I be removed from the research without my OK?

You will not be withdrawn from the study without your direct consent.

### What else do I need to know?

This research is being funded by **National Institute of Diabetes and Digestive and Kidney Diseases** (NIDDK).

If you agree to take part in this research study, you will receive a \$25 honorarium for your time and effort. This amount will not be pro-rated as you will receive the full payment for the completion of the interview.

Private, identifiable information will only be used for research and statistical purposes. However, if you indicate future criminal intent, elder abuse, child abuse, or plans to harm self or others, the researchers are required by law to report this to the authorities.

Project findings and reports prepared for dissemination will not contain information that can reasonably be expected to be identifiable.

Total payments within one calendar year that exceed \$600 will require the University to report these payments annually to the IRS and you. This may require you to claim the compensation you receive for participation in this study as taxable income. VCU is required by federal law to collect your social security number. Your social security number will be kept confidential and will only be used to process payment.

Please be aware that the investigative team and the University may receive money for the conduct of this study.

# **Signature Block for Capable Adult**

| Your signature documents your permission to take part in this rese | arch. | |
|---|---|---|
| Signature of subject | Date | |
| Printed name of subject | Date | |
| Signature of person obtaining consent | Date | |
| Printed name of person obtaining consent | | |
| [Add the following block if a witness will observe the conse<br>documentation or illiterate se | | consent |
| My signature below documents that the information in the consent was accurately explained to, and apparently understood by, the su the subject. | • | |
| Signature of witness to consent process | Date | |
| Printed name of person witnessing consent process | <br>Date | |

# Permission to Take Part in a Human Research Study

ICF version number: Version 1

Title of research study¹: Using Grassroots Wellness Coaching to Enhance Reach and Sustainability of Behavioral Weight Management

Investigator: Maghboeba Mosavel, PhD, Professor: (804) 628-2929 and Jessica G. LaRose, PhD,

Professor: (804) 628-7521

<u>Key Information</u>: The following is a short summary of this study to help you decide whether or not to be a part of this study. More detailed information is listed later on in this form.

# Why am I being invited to take part in a research study?

We invite you to take part in a research study because:

- You are a community Stakeholder, or
- Your organization has been identified as involved in a health and wellness initiative in Petersburg.

# What should I know about a research study?

- Someone will explain this research study to you.
- Whether or not you take part is up to you.
- You can choose not to take part.
- You can agree to take part and later change your mind.
- Your decision will not be held against you.
- You can ask all the questions you want before you decide.

# Why is this research being done?

This research is being conducted as part of the WE 2.0 Project, which has been active in Petersburg for many years. In this program, local residents were trained to be group leaders, and they invited their family, friends, and acquaintances to join. As part of the program, a variety of materials were developed based on feedback and input from the Petersburg community. These materials include a walking club toolkit, videos, infographics, a website, and other health and wellness content.

The purpose of this study is to find out how these materials might be helpful to organizations or others in the community. Specifically, we aim to share the tools and materials developed, learn whether organizations and the people they serve might find them useful, and hear suggestions or recommendations for slight adjustments to make them more broadly applicable. Additionally, the research seeks to understand how aspects of the 12-week health and wellness program that we completed with a small group could now benefit the larger community. As researchers, we want to understand how the materials that we developed in the WE project can benefit others.

# How long will the research last and what will I need to do?

You will be asked to participate in a one-time, 45-minute Zoom meeting with one member of the WE research team to share insights on your organization and provide feedback on the materials that will be shared with


<sup>&</sup>lt;sup>1</sup> This template satisfies AAHRPP elements I.1.G, I.4.A, I-9, II.3.C-II.3.C.1, II.3.E, II.3.F, II.4.B, III.1.F, III.1.G

other communities. Only the audio portion of this meeting will be downloaded and analyzed for the results. There are no additional tasks to be completed once you finish.

More detailed information about the study procedures can be found under "What happens if I say yes, I want to be in this research?"

# Is there any way being in this study could be bad for me?

This study is considered low risk. You won't face any physical harm or emotional distress, and we've designed everything to respect your privacy and make sure you feel comfortable and at ease throughout the process.

We do understand that this meeting might feel a little uncomfortable. If that happens, we want you to know those feelings are normal and should only be short-term. To help, we'll create a supportive, judgment-free space during the interviews. This study is all about hearing from you and how you think the information we developed could be useful to Petersburg residents and/or organizations. You may think they cannot be useful or they can be useful - there is no right or wrong answer.

# Will being in this study help me in any way?

We cannot promise any direct benefits to you from being part of this research. However, possible benefits include the opportunity to share your experiences and insights, which may help improve wellness programs in your community.

Your experiences and insights can possibly help improve the program to make it more beneficial for others in Petersburg or communities outside of Petersburg.

# What happens if I do not want to be in this research?

Participation in research is completely voluntary. You can decide to participate, not participate, or discontinue participation at any time without penalty or loss of benefits to which you are otherwise entitled.

Your alternative to participating in this research study is to not participate.

<u>Detailed Information</u>: The following is more detailed information about this study in addition to the information listed above.

#### Who can I talk to?

If you have questions, concerns, or complaints, or think the research has hurt you, talk to the research team at (804) 396-4556 or send us an email: WEPetersburg2.0@vcuhealth.org.

This research has been reviewed and approved by an Institutional Review Board ("IRB"). You may talk to them at (804) 828-0868 or HRPP@vcu.edu if:

- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.
- You want to talk to someone besides the research team.
- You have questions about your rights as a research subject.
- You want to get information or provide input about this research.

# How many people will be studied?

We expect about 40 people to take part in this research study out of 50 people in the entire study

# What happens if I say yes, I want to be in this research?

If you agree to participate in this study, you will be asked to complete a one-time, 45 minute Zoom audio meeting with a member of the WE 2.0 Project research team. This interview will be scheduled at a time that is most convenient for you.

# What are my responsibilities if I take part in this research?

During this meeting, you will be responsible for providing your personal insights about various aspects of the WE 2.0 and offer any suggestions that could improve this study for other communities in the future.

As a stakeholder, you will also have the option to choose whether or not you would like to disclose your identity and the organization that you represent.

# What happens if I say yes, but I change my mind later?

You can leave the research at any time; it will not be held against you. If you choose to withdraw for any reason, all data collected will be carefully disposed of to eliminate any risk of personal information being misused. In addition, you will not be withdrawn from the study without your explicit consent.

All data that is collected will be used for research purposes only. Your data will be identified by an ID number and safely stored in our database. Access to all data will be limited to study personnel.

We will do our best to protect your data during storage and when it is shared. You have the option to choose whether your identity and the identity of your organization will be shared or remain anonymous. However, there remains a possibility that someone could identify you, even if you choose to remain anonymous. While we take all reasonable measures to ensure your privacy, we cannot eliminate all risks.

# What happens to the information collected for the research?

Efforts will be made to limit the use and disclosure of your personal information, including research study and medical records, to people who have a need to review this information. We cannot promise complete secrecy. Organizations that may inspect and copy your information include the IRB and other representatives of this organization.

# Will my data or samples be used for future research?

Your information collected as part of this research will not be used or distributed for future research studies, even if all of your identifiers are removed.

# Can I be removed from the research without my OK?

You will not be withdrawn from the study without your explicit consent.

### What else do I need to know?

# This research is being funded by *National Institute of Diabetes and Digestive and Kidney Diseases* (*NIDDK*)

If you agree to take part in this research study, you will receive a \$25 honorarium for your time and effort. This amount will not be pro-rated as you will receive the full payment based upon completion of this one time meeting.

Private, identifiable information will only be used for research and statistical purposes. However, if you indicate future criminal intent, the researchers are required by law to report this to the authorities.

Project findings and reports prepared for dissemination will not contain information that can reasonably be expected to be identifiable.


Total payments within one calendar year that exceed \$600 will require the University to report these payments annually to the IRS and you. This may require you to claim the compensation you receive for participation in this study as taxable income. VCU is required by federal law to collect your social security number. Your social security number will be kept confidential and will only be used to process payment.

Please be aware that the investigative team and the University may receive money for the conduct of this study.

# Consent to Share your Information

- I provide permission to have my identity, role, and that of my organization known in the reporting of the results
- I DO NOT provide permission to have my identity, role, and that of my organization known in the reporting of the results

# **Signature Block for Capable Adult**

Your signature documents your permission to take part in this research.

| Signature of subject | Date | |
|---|---|---|
| Printed name of subject | Date | |
| Signature of person obtaining consent | Date | |
| Printed name of person obtaining consent | | |
| [Add the following block if a witness will observe the condition of illiteration or illiterati | • | of consent |
| My signature below documents that the information in the conwas accurately explained to, and apparently understood by, the subject. | • | |
| Signature of witness to consent process | Date | Page 4 of |

| 1/9/2025 |
|-------------|
| IRB on |
| VCU |
| by the |
| Approved by |